CLINICAL TRIAL: NCT00984165
Title: Pilot Study of Radiation-Enhanced Allogeneic Cell Therapy for Progressive Hematologic Malignancy After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual, PI left NIH and primary endpoint not met.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090224; 09-C-0224
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-03

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemias; Multiple Myeloma With Plasmacytoma
Keywords: Allotransplant; Relapse; Radiation; Donor Lymphocyte Infusion; Hematologic Malignancies; Multiple Myeloma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Hematologic Neoplasms; Multiple Myeloma | interventions — Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Donor Lymphocyte Infusion/Radiation (Experimental): Subjects will receive a unmanipulated donor lymphocyte infusion (DLI) on Day 1 after radiation (single, 8-Gy fraction to the maximum number of lesions).
  Interventions: Procedure: Single fraction radiation; Biological: Donor Lymphocyte Infusion (DLI)
- Radiation/No Donor Lymphocyte Infusion (Active Comparator): Subjects will receive radiation (single, 8-Gy fraction to the maximum number of lesions).
  Interventions: Procedure: Single fraction radiation
- Donor Lymphocyte Infusion - Control (Active Comparator): Subjects will receive a unmanipulated donor lymphocyte infusion (DLI) on Day 0.
  Interventions: Biological: Donor Lymphocyte Infusion (DLI)
- Donor Lymphocyte Infusion - Donor (Active Comparator): Healthy subjects who donated lymphocytes for infusion on a treatment Arm.
  Interventions: Procedure: Apheresis

INTERVENTIONS:
Procedure: Single fraction radiation — 8-Gy fraction of radiation
  Arms: Donor Lymphocyte Infusion/Radiation; Radiation/No Donor Lymphocyte Infusion
Biological: Donor Lymphocyte Infusion (DLI) — Unmanipulated Donor Lymphocyte Infusion
  Arms: Donor Lymphocyte Infusion - Control; Donor Lymphocyte Infusion/Radiation
Procedure: Apheresis — Donors will undergo a 5-liter apheresis procedure on a CS-3000 or equivalent machine.
  Arms: Donor Lymphocyte Infusion - Donor

SUMMARY:
Background:

* Allogeneic hematopoietic stem cell transplantation (allotransplant) has been used to treat many kinds of cancer that develop in cells from the blood or immune system. After allotransplant, donor cells take over production of the recipient s blood and immune cells, and donor immune cells can directly attack and control tumor. However, for cancers that do not respond to allotransplant, there are no proven cures.
* A single treatment with radiation can improve the potency of immune-cell therapies. This is probably because the tumor tissue is damaged in a way that new tumor proteins are exposed, attracting immune cells to the tumor. By giving only a single dose of radiation, the immune cells that are attracted to the tumor are allowed to survive and function in their usual way, traveling throughout the body and educating other immune cells to recognize tumor, and to activate and expand in order to kill the tumor cells. Some research has shown that radiation may have a widespread effect on stimulating the immune system, educating immune cells to recognize and control tumors that have not been radiated.

Objectives:

- To determine whether a single treatment of radiation will help donor immune cells control cancer after allotransplant without causing excessive side effects.

Eligibility:

* Recipients: Individuals 18 years of age and older who have blood cancers that have not responded to allotransplant.
* Donors: Healthy individuals 18 years of age and older who were previous allotransplant donors for one of the study recipients.

Design:

* Donors will provide additional blood immune cells, called lymphocytes, through apheresis. Apheresis involves drawing blood, separating out the lymphocytes, and returning the rest of the blood to the donor.
* Recipients will receive a single dose of radiation to the greatest amount of tumor that can be irradiated safely. Researchers will intentionally leave some tumor that will not be radiated in order to evaluate whether there is a widespread response to the treatment.
* There are two treatment arms on the study.
* Arm 1: Study participants who have donor lymphocytes available and who have not had major complications from the allotransplant will be given a dose of donor cells after they receive radiation, to provide an additional boost to the donor immune response.
* Arm 2: Study participants who cannot receive donor lymphocytes because their donor is not available, they received an allotransplant from a partially matched relative, or they have had significant complications from the allotransplant - will receive radiation without additional donor lymphocytes.
* All recipients will be followed closely for side effects and for tumor response to radiation with or without donor lymphocytes. Additional tests will be performed, including tumor biopsies, bone marrow samples, and blood draws, in order to study the immune effects of radiation and donor lymphocytes.
* A separate, control group of allotransplant recipients will not receive radiation. This group will include participants whose transplant doctors plan to use donor lymphocyte therapy alone to control cancer progression. This group will donate blood immune cells through blood draws and apheresis. These cells will be examined to study the immune effects of receiving donor lymphocytes without radiation.

DETAILED DESCRIPTION:
Background:

* The prognosis for patients with cancer who have relapsed or progressive disease after allogeneic hematopoietic stem cell transplantation (allotransplant) is poor. Effective therapies for patients who fail withdrawal of immune suppression and administration of donor lymphocyte infusions (DLI) have not been identified.
* Increasing the efficacy of allotransplant without increasing toxicity is a major goal of transplantation research. A major research effort within the Experimental Transplantation and Immunobiology Branch (ETIB) is to identify ways to build on the allogeneic platform to treat relapse after allotransplant.
* We hypothesize that a single fraction of radiation to tumor prior to administration of donor lymphocytes will increase the potency of systemic graft-versus-tumor (GVT) effects without increasing graft-versus-host disease (GVHD).

Objectives:

- To determine the safety, in relation to GVHD and allograft function, and efficacy, in terms of systemic tumor response, of administering single-fraction, targeted radiotherapy with or without DLI to patients with persistent tumor after allotransplant.

Eligibility:

* Adults with hematologic malignancies that progress or recur after allotransplant, successful donor T cell engraftment, and trial of withdrawal of immune suppression.
* Disease that is amenable to radiation as well as additional measurable disease outside the radiation field.
* Subjects with treatment-refractory acute or chronic GVHD will not be eligible.

Design:

* Subjects will receive radiation in a single, 8-Gy fraction to sites of disease. At least one site of measurable disease will remain untreated with radiation for evaluation of systemic response.
* There will be two arms. Arm A will include subjects with available donor lymphocytes and who have not had GVHD requiring systemic treatment; they shall receive a DLI the day after completion of radiation. Arm B will include those who have previously required systemic therapy for GVHD, are at high risk of significant GVHD, and/or who do not have available donor lymphocytes; they shall receive radiation without DLI.
* Additional disease that is outside the field of radiation will be monitored for systemic effects of the therapy.
* Subjects will be monitored on an outpatient basis for the development or exacerbation of GVHD, excessive hematologic toxicity or other toxicity from radiation, and for tumor responses for at least 60 days.
* Enrollment:

  * Treatment Subjects: The protocol will treat 21 subjects per arm (total 42). There are stopping rules after 8 and 15 patients per arm for excessive GVHD or radiation toxicity.
  * DLI Control Subjects; 15 control subjects who receive DLI for persistent disease as part of their care on another National Institutes of Health (NIH) protocol, will be included to compare the immunologic effects of radiation followed by DLI (Arm A) with DLI alone.
  * Donor Subjects: Related donors of Arm A Treatment Subjects and DLI Control Subjects will be enrolled for collection of clinical DLI product, a portion of which will be used for research (up to 36 Donor Subjects).

ELIGIBILITY:
* INCLUSION CRITERIA:

Treatment Subjects:

* Patients must have received allotransplant (related or unrelated donor) for hematologic malignancies and have disease progression with a component of solid-phase disease. Eligible diagnoses will include any acute or chronic leukemia with a solid-phase component, Hodgkin's lymphoma, any non-Hodgkin's lymphoma, including mantle cell lymphoma, multiple myeloma. Pathology slides from patients pretransplant diagnoses will be reviewed by National Cancer Institute (NCI)/Center for Cancer Research (CCR) Department of Pathology.
* Patients must have at least two distinct sites of disease:
* At least one site must be in solid phase and amenable to irradiation, determined by Radiation Oncology evaluation.
* In addition to the target(s) of irradiation, there must be disease that is discrete from local effects of the radiation that can be evaluated for systemic response to therapy.
* Patients must have disease that has failed to respond after a minimum of four weeks to:
* Evidence of complete donor-T cell engraftment (greater than 90% chimerism) of the circulating T cells
* A trial of tapering immunosuppressive therapy, including trials that are discontinued due to development or flare of graft versus host disease (GVHD)
* Patients must be 18 - 75 years of age.
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 3 (Karnofsky greater than or equal to 50%).
* Life expectancy greater than or equal to 1 month.

Arm A

* Patients with minimal to no clinical evidence of acute GVHD (Grade 0-I) or mild- chronic GVHD (GVHD Score of no more than 1 in no more than two organ systems) while off of systemic immunosuppressive therapy.
* Available source of clinical donor lymphocyte cell product, including stem cell-mobilized product.
* Patients whose related allotransplant donor is available, eligible and enrolled on this or another National Institutes of Health (NIH)/Clinical Center (CC) protocol that permits collection of a clinical donor lymphocyte cell product, and donors are first-degree relatives with genotypic identity at 5-6/6 human leukocyte antigen (HLA) loci (HLA- A, B, and DR. Haploidentical (less than 5/6 genotypic identity) allotransplant recipients will not be eligible, due to risk of severe GVHD with donor lymphocyte infusion (DLI).
* Patients whose related or unrelated allotransplant donors are unavailable or ineligible, but who have cryopreserved donor lymphocyte cell products available for use on this trial.

Arm B

* Patients with history of GVHD. Specifically:

  * Patients who have a past history of resolved grade III acute GVHD or moderate/severe chronic GVHD and who are no longer requiring systemic therapy to treat GVHD.
  * Patients who require continued prophylaxis with steroid-sparing agents, e.g., cyclosporine. Due to concerns that sirolimus (rapamycin) could interfere with the potential efficacy of radiation-enhanced allogeneic cell therapy, patients on sirolimus as part of GVHD control must be switched to another agent two weeks prior to enrollment.
  * Patients with GVHD controlled with local therapy, e.g., topical steroids, budesonide.
  * Patients with controlled acute GVHD (Grade I-III) or chronic-moderate/severe GVHD on a stable (at least four weeks) or tapering dose of systemic immunosuppression will be eligible for enrollment.
* Patients who do not have donor lymphocytes available for use on this trial, including recipients of unrelated donor allografts.
* Patients whose allotransplant was from a haploidentical (less than 5/6 genotypic identity) related donor.
* Provision for a Durable Power of Attorney.
* Ability to give informed consent.

Donor Subjects:

* Donors are the same individual whose cells were used as the source for the enrolling Arm A Treatment Subject or DLI Control Subjects original allotransplant.
* Age 18 - 90.
* Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.
* Donors must be human immunodeficiency virus (HIV) negative, hepatitis B surface antigen negative, and hepatitis C antibody negative.

DLI Control Subjects:

The DLI Control Subjects will serve as a comparison for Arm A, and eligibility criteria are intended to enroll subjects who are similar with respect to allotransplant characteristics.

* Patients must be 18-75 years of age.
* Patients who have received an allotransplant to treat malignancy and who are going to receive an unmanipulated or stem-cell mobilized DLI to treat persistent tumor as part of their treatment program on another National Institutes of Health (NIH)/Clinical Center (CC) protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 3 (Karnofsky performance status of greater than or equal to 50%).
* Life expectancy greater than or equal to 1 month.
* Patients with minimal to no clinical evidence of acute GVHD (Grade 0-I) or mild- chronic GVHD while off of systemic immunosuppressive therapy.
* Available source of clinical donor lymphocyte cell product, including a stem cell-mobilized product.

  * Patients whose related allotransplant donor is available, eligible and enrolled on this or another NIH/CC protocol that permits collection of a clinical donor lymphocyte cell product, and donors are first-degree relatives with genotypic identity at 5-6/6 human leukocyte antigen (HLA) loci (HLA- A, B, and DR. Haploidentical (less than 5/6 genotypic identity) allotransplant recipients will not be eligible, for consistency with Arm A Subjects.
  * Patients whose related or unrelated allotransplant donors are unavailable or ineligible, but who have cryopreserved donor lymphocyte cell products available for clinical use on this trial.
* Patients must have disease that has failed to respond after a minimum of four weeks to:
* Evidence of complete donor-T cell engraftment (greater than 90% chimerism) of the circulating T cells.
* A trial of tapering immunosuppressive therapy, including trials that are discontinued due to development or flare of GVHD.
* Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis or consent to a large-volume (70cc) blood draw.
* Permission from their treating transplant physician or designee to participate on study.
* Ability to give informed consent.

EXCLUSION CRITERIA:

Treatment Subjects:

* Tumor-directed therapy within two weeks of DLI.
* Patients with rapid disease progression or aggressive tumor histology which, in the opinion of the principal investigator (PI), is likely to require urgent therapy within 60 days in order to preserve organ function or quality of life, and there is an available standard therapy to which the patient has a reasonable chance of responding.
* Progressive disease that, in the opinion of the PI, requires urgent standard therapy, e.g., threatened organ function, acceptable quality of life, etc.
* Uncontrolled GVHD, i.e., either acute GVHD Grade III or chronic-moderate/severe GVHD that has not responded to the current dose of systemic therapy or any history of steroid-refractory acute GVHD, Grade IV acute GVHD, or chronic-severe GVHD.
* Active infection that is not responding to antimicrobial therapy.
* Active psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent (as determined by Principal Investigator and/or her designee).
* Pregnant or lactating. Subjects of childbearing potential must use an effective method of contraception. The effects of the immunosuppressive medications that could be required to treat GHVD are likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to an infant.
* Absolute neutrophil count of less than 500 cells/microL. At the PIs discretion, patients with marrow replacement by tumor as the probable etiology of an absolute neutrophil count of less than 500 cells/microL may be eligible for enrollment.
* In order to prevent delay of potentially stabilizing palliative therapy, the following conditions will exclude eligibility: untreated active leptomeningeal involvement with malignancy, untreated brain metastasis, and other organ-threatening diseases in which palliative treatment options with reasonable probability of efficacy (15% or higher) are available. Patients with these conditions for whom available palliative options have been tried or deemed unacceptable but who otherwise meet eligibility criteria may, at the discretion of the PI, be considered for enrollment.

Donor Subjects:

* History of a psychiatric disorder that the PI determines might compromise compliance with transplant protocol, or that does not allow for appropriate informed consent.
* Hypertension that is not controlled by medication, history of stroke, or severe heart disease (donors with symptomatic angina will be excluded). Donors with a history of coronary artery bypass grafting or angioplasty who are symptom free will receive a cardiology evaluation and be considered on a case-by-case basis.
* History of prior malignancy. However, cancer survivors who have undergone potentially curative therapy and have had no evidence of that disease for at least 5 years may be considered for lymphocyte donation on a case-by-case basis.
* Anemia (hemoglobin (Hb) less than 11 gm/dl) or thrombocytopenia (platelets less than 100,000 per ml). However, potential donors with Hb levels less than 11 gm/dl that is due to iron deficiency will be eligible as long as the donor is initiated on iron replacement therapy and the case is individually approved by NIH Department of Transfusion Medicine (DTM).
* Pregnancy. Donor Subjects of childbearing potential must use an effective method of contraception until after completion of apheresis. The effects of apheresis are unknown to be safe to a fetus.

DLI Control Subjects:

* Tumor-directed therapy within two weeks of DLI.
* Uncontrolled GVHD
* Pregnant or lactating. Subjects of childbearing potential must use an effective method of contraception until after completion of apheresis. The effects of apheresis are unknown to be safe to a fetus.
* History of a psychiatric disorder that the PI determines might compromise compliance with protocol, or that does not allow for appropriate informed consent.
* Hypertension that is not controlled by medication, history of stroke, or severe heart disease (subjects with symptomatic angina will be excluded).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2013-01-18 (Actual); Study Completion 2013-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wattenberg MM, Kwilas AR, Gameiro SR, Dicker AP, Hodge JW. Expanding the use of monoclonal antibody therapy of cancer by using ionising radiation to upregulate antibody targets. Br J Cancer. 2014 Mar 18;110(6):1472-80. doi: 10.1038/bjc.2014.79. Epub 2014 Feb 20. PMID 24556625
- [Background] Hasumi K, Aoki Y, Wantanabe R, Mann DL. Clinical response of advanced cancer patients to cellular immunotherapy and intensity-modulated radiation therapy. Oncoimmunology. 2013 Oct 1;2(10):e26381. doi: 10.4161/onci.26381. Epub 2013 Oct 17. PMID 24349874
- [Background] Schirrmacher V. Complete remission of cancer in late-stage disease by radiation and transfer of allogeneic MHC-matched immune T cells: lessons from GvL studies in animals. Cancer Immunol Immunother. 2014 Jun;63(6):535-43. doi: 10.1007/s00262-014-1530-2. Epub 2014 Mar 9. PMID 24610041
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0224.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donor Lymphocyte Infusion/Radiation | Radiation/No Donor Lymphocyte Infusion | Donor Lymphocyte Infusion - Control | Donor Lymphocyte Infusion - Donor
Started | 9 | 1 | 4 | 4
Completed | 2 | 0 | 4 | 0
Not Completed | 7 | 1 | 0 | 4
Not completed — Death on study | 2 | 0 | 0 | 0
Not completed — Disease progression on study | 5 | 1 | 0 | 0
Not completed — Death of recipient | 0 | 0 | 0 | 1
Not completed — New protocol | 0 | 0 | 0 | 1
Not completed — P+/donor pair removed from protocol | 0 | 0 | 0 | 1
Not completed — removed with a pair recipient | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donor Lymphocyte Infusion/Radiation | Radiation/No Donor Lymphocyte Infusion | Donor Lymphocyte Infusion - Control | Donor Lymphocyte Infusion - Donor | Total
Number analyzed (Participants) | 9 | 1 | 4 | 4 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 4 | 4 | 17
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.78 (14.84) | 33.5 (0) | 29.5 (3.41) | 34.83 (3.97) | 36.15 (0.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 3 | 8
  Male | 6 | 1 | 2 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 1 | 4 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 1 | 4 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 1 | 4 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Response to Graft Versus Host Disease (GVHD) Treatment
Description: The following criteria is used to determine response to GVHD treatment. Complete response (CR) is complete resolution of all clinical signs and symptoms of acute GVHD. Partial response (PR) is 50% reduction in skin rash, stool volume or frequency, and/or total bilirubin. Failure to maintain adequate performance status (Karnofsky Score >/= 70%). Non-responder (NR) <50% reduction in skin rash, stool volume or frequency, and/or total bilirubin. Failure to maintain adequate performance status (Karnofsky Score </= 70%). Progressive disease (PD) is further progression of signs and symptoms of acute GVHD, and/or decline in performance status after the initiation of therapy.
Time Frame: Up to 100 days
Population: No results were collected on the Donor Lymphocyte Infusion-Donor "Arm". This arm allowed for collection of the lymphocytes on healthy donors for infusion on the DLI/Radiation Arm or the DLI/Control Group.
Measure: Number; unit: participants
Groups:
- Donor Lymphocyte Infusion-Control: Subjects will receive a unmanipulated donor lymphocyte infusion (DLI) on Day 0.
Arm/Group | Donor Lymphocyte Infusion/Radiation | Radiation/No Donor Lymphocyte Infusion | Donor Lymphocyte Infusion-Control
Number analyzed (Participants) | 9 | 1 | 4
participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 1 | 0 | 0
  Non-responder (NR) | 6 | 1 | 3
  Progressive Disease (PD) | 2 | 0 | 1

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Lymphocyte Infusion/Radiation | Radiation/No Donor Lymphocyte Infusion | Donor Lymphocyte Infusion - Control | Donor Lymphocyte Infusion - Donor
Number analyzed (Participants) | 9 | 1 | 4 | 4
Participants | 9 | 1 | 4 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 36 months.
Arm/Group | Donor Lymphocyte Infusion/Radiation | Radiation/No Donor Lymphocyte Infusion | Donor Lymphocyte Infusion - Control | Donor Lymphocyte Infusion - Donor
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/1 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/9 | 0/1 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 9/9 | 1/1 | 4/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor Lymphocyte Infusion/Radiation (N=9) | Radiation/No Donor Lymphocyte Infusion (N=1) | Donor Lymphocyte Infusion - Control (N=4) | Donor Lymphocyte Infusion - Donor (N=4)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (coma) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (aspergillis (+) in sputum) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (sputum, pseudomonas (+)) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor Lymphocyte Infusion/Radiation (N=9) | Radiation/No Donor Lymphocyte Infusion (N=1) | Donor Lymphocyte Infusion - Control (N=4) | Donor Lymphocyte Infusion - Donor (N=4)
Activated partial thromboplastin time prolonged (Investigations) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (10) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (b/l ear fullness) (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haptoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (7) | 1 (1) | 1 (2) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (17) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (9) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 6 (14) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (angular cheilitis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2014-02-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT00984165/Prot_000.pdf
  • Informed Consent Form: DLI Control consent (2011-12-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT00984165/ICF_001.pdf
  • Informed Consent Form: Recipient consent (2011-12-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT00984165/ICF_002.pdf
  • Informed Consent Form: Donor consent (2011-12-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT00984165/ICF_003.pdf